CLINICAL TRIAL: NCT03284216
Title: The Effects of Hyperglycemia on the Response to Acute Exercise.
Brief Title: Hyperglycemia and Exercise.
Acronym: GlucotoxEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ERN_16-0193
Record Dates: First submitted 2017-02-28; First posted 2017-09-15 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Aerobic Exercise; Hyperglycemia; Glucose Metabolism Disorders (Including Diabetes Mellitus)
MeSH Terms: conditions — Hyperglycemia; Glucose Metabolism Disorders | interventions — Pharmaceutical Preparations; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal glycemia + exercise (Other): Participants will be studied in the fasting state under normal blood glucose conditions whereby no glucose will be administered, but an exercise bout will be completed.
  Interventions: Behavioral: Exercise
- Steady-state hyperglycemia + exercise (Experimental): Participants will be studied during experimental steady-state hyperglycemia-induced via a variable-rate intravenous glucose infusion, and an exercise bout will be completed.
  Interventions: Procedure: Steady-state hyperglycemia; Behavioral: Exercise
- Fluctuating hyperglycemia + exercise (Experimental): Participants will be studied during experimental fluctuating hyperglycemia-induced via repeated intravenous glucose injections, and an exercise bout will be completed.
  Interventions: Procedure: Fluctuating hyperglycemia; Behavioral: Exercise
- Normal glycemia, no exercise (No Intervention): Participants will be studied in the fasting state under normal blood glucose conditions whereby no glucose will be administered and no exercise will be completed.

INTERVENTIONS:
Procedure: Steady-state hyperglycemia — Experimental "diabetic like" steady-state hyperglycemia will be induced via a continuous-rate intravenous glucose infusion.
  Other Names: Drug (metabolite infusion)
  Arms: Steady-state hyperglycemia + exercise
Procedure: Fluctuating hyperglycemia — Experimental "diabetic like" fluctuating hyperglycemia will be induced via repeated intravenous glucose injections.
  Other Names: Drug (metabolite injection)
  Arms: Fluctuating hyperglycemia + exercise
Behavioral: Exercise — Moderate-intensity exercise bout (45-minutes of cycling at 70% of their heart rate max) at T=4.5 hours
  Arms: Fluctuating hyperglycemia + exercise; Normal glycemia + exercise; Steady-state hyperglycemia + exercise

SUMMARY:
This study will determine whether exposure to short-term high blood glucose levels impairs exercise-induced adaptations in glucose tolerance, and whether the pattern of high blood glucose levels plays a role.

DETAILED DESCRIPTION:
Healthy male volunteers will undergo a screening visit and four experimental trials.

Screening Visit: Having read the participant info sheet, a study investigator will discuss the project with the potential participant who will have the chance to ask any questions. Informed consent will be sought and a General Health Questionnaire will be completed. Body weight, height, and skinfold measurements will be taken. Participants will also complete an exercise test to measure V̇O2max test along with heart rate and blood pressure measurements.

Individuals eligible for inclusion in the study will then return to the lab for four experimental trials, each separated by ~1 week. Trials will be completed using a randomised, counter-balanced, cross-over design. Between experimental trials, participants will be instructed to maintain their normal diet and activity habits. During the 48 hours prior to each experimental trial participants will be instructed to refrain from vigorous exercise and alcohol. For 3 days prior to each experimental trial, participants will record their dietary intake, and wear an accelerometer and a continuous glucose monitor to measure physical activity levels and glucose control.

Experimental Trials: Participants will arrive at the laboratory in the morning (~8 am) following an overnight (~10 hour) fast from food and drink (except water) since 10pm the previous evening. Upon entering the laboratory, body composition (height, weight, waist circumference) will be assessed and a cannula will be placed into a vein in each arm (one for infusion of glucose, one for blood sampling). Resting cardiovascular measures (heart rate, blood pressure, oxygen saturation) will be collected followed by an assessment of cognitive function followed immediately by one of the four 3.5 hour interventions:

* Trial A (normoglycaemia prior to exercise): This will involve no glycaemic intervention and the participant will remain in a rested, normoglycaemic state throughout all subsequent procedures.
* Trial B (steady hyperglycaemia prior to exercise): This will involve a continuous constant-rate glucose infusion to establish a steady hyperglycaemic profile. Specifically, 1.2g/kg glucose will be infused at a constant infusion rate across 3.5 hrs (equivalent to 5.71 mg/kg/min).
* Trial C (fluctuating hyperglycaemia prior to exercise): This will involve repeated glucose injections so as to cause multiple fluctuations in glycaemia. Specifically, 1.2 g/kg glucose will be infused via 8 equal boluses every 30 minutes across 3.5 hrs (the equivalent of 0.15 g/kg per bolus infused over 3.5 minutes at a rate of 42.86 mg/kg/min) interspersed with periods of no infusion.
* Trial D (normoglycaemia, no exercise): This will be identical to trial A, except there will be no exercise bout.

After 3.5 hours, the above-described glycaemic intervention will stop, and be followed immediately by the collection of post-intervention blood samples, assessment of cardiovascular response and assessment of cognitive function. Participants will then complete an exercise bout consisting of 45 minutes of moderate intensity (70% HRmax) continuous cycling, during which energy expenditure will be measured by indirect calorimetry. Post-exercise blood samples will be collected, and catheters will be removed. Participants will be fed a meal. Before leaving the lab, they will also be provided with an evening meal to be consumed at home at 7 pm, and a breakfast and lunch meal for the following day (to be consumed at 7 am and 12 pm, respectively). Participants will then return to the laboratory for 5 minutes the afternoon after the trial day (~3 pm) to remove the accelerometer and continuous glucose monitor, marking the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged between 18 and 50 years.
* Body Mass Index of between 19 and 30 kg/m2.

Exclusion Criteria:

* Smoking.
* Regularly use of anti-inflammatory medication.
* More than 2 kg weight change in the last 6 months, and/or have undergone weight loss surgery.
* Previous or current cancer or chronic haematological, pulmonary, cardiac, hepatic, renal, metabolic, or gastrointestinal diseases.
* Currently engaged in moderate or vigorous exercise on more than 5 days per week.
* Contraindication to exercise.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-08 (Actual)

PRIMARY OUTCOMES:
Exercise-induced change in blood glucose control. | In all trials, glucose control will be determined between the time-point immediately after exercise and 24 hours after exercise.
  In all trials, continuous glucose monitoring (CGM) will be used to assess the change in glucose control compared to baseline for 24 hours after-exercise, under diet-controlled but otherwise free-living conditions.

SECONDARY OUTCOMES:
Hyperglycemia-induced change in inflammation. | In all trials, inflammation will be determined at baseline (T=0 hours) and at T=3.5 hours. The glycemic interventions take place between baseline (T=0 hours) and T=3.5 hours.
  In all trials, plasma cytokine levels (IL-6, TNF-alpha, IL-1ra) will be measured at baseline (T=0 hours) and immediately after each glycaemic intervention (T=3.5 hours). The interventions will take place between baseline (T=0 hours) and T=3.5 hours.
Hyperglycemia-induced change in cognitive function. | In all trials, cognitive function will be determined at baseline (T=0 hours) and at T=3.5 hours. The glycemic interventions take place between baseline (T=0 hours) and T=3.5 hours.
  In all trials, cognitive function tests (CANTAB) to measure executive functioning and verbal memory will be administered at baseline (T=0 hours) and immediately after each glycaemic intervention (T=3.5 hours). The interventions will take place between baseline (T=0 hours) and T=3.5 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Solomon TPJ, Carter S, Haus JM, Karstoft K, von Holstein-Rathlou S, Nielsen MS, Gillum MP. Plasma FGF21 concentrations are regulated by glucose independently of insulin and GLP-1 in lean, healthy humans. PeerJ. 2022 Jan 19;10:e12755. doi: 10.7717/peerj.12755. eCollection 2022. PMID 35111398
- [Derived] Carter S, Solomon TPJ. Exercise-Induced Improvements in Postprandial Glucose Response Are Blunted by Pre-Exercise Hyperglycemia: A Randomized Crossover Trial in Healthy Individuals. Front Endocrinol (Lausanne). 2020 Oct 15;11:566548. doi: 10.3389/fendo.2020.566548. eCollection 2020. PMID 33178135